CLINICAL TRIAL: NCT04081350
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Multiple-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Subcutaneous LY3471851 in Patients With Atopic Dermatitis
Brief Title: A Study of LY3471851 in Participants With Eczema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17240; J1P-MC-KFAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02-15

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10 µg/kg LY3471851 (Active Comparator): Participants received subcutaneous (SC) injection of 10 microgram per kilogram (μg/kg) LY3471851 every 2 weeks for a treatment period of 12 weeks.
  Interventions: Drug: LY3471851
- 12 µg/kg LY3471851 (Active Comparator): Participants received subcutaneous injection of 12 μg/kg LY3471851 every 2 weeks for a treatment period of 12 weeks.
  Interventions: Drug: LY3471851
- 24 µg/kg LY3471851 (Active Comparator): Participants received subcutaneous injection of 24 μg/kg LY3471851 every 2 weeks for a treatment period of 12 weeks.
  Interventions: Drug: LY3471851
- Placebo (Placebo Comparator): Participants received subcutaneous injection of placebo every 2 weeks for a treatment period of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3471851 — Administered SC
  Other Names: NKTR-358
  Arms: 10 µg/kg LY3471851; 12 µg/kg LY3471851; 24 µg/kg LY3471851
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about the safety and side effects of LY3471851 when given by injection just under the skin to participants with eczema. The study will last up to 48 weeks and may include up to 23 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of atopic dermatitis (AD) for least 12 months
* Have active AD according to study specific criteria
* Be willing and able to undergo skin biopsies

Exclusion Criteria:

* Have received certain topical medications for AD within 14 days prior to baseline
* Have received certain systemic medications for AD within 4 weeks prior to baseline
* Have received LY3471851 previously

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Study Completion (up to Week 48)
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3471851 | Postdose on Day 1 through Day 14
  PK: AUC of LY3471851
PK: Trough Concentrations (Ctrough) of LY3471851 | Week 12
  PK: Ctrough of LY3471851
PK: Maximum Concentration (Cmax) of LY3471851 | Postdose on Day 1 through Day 14
  PK: Cmax of LY3471851

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (20):
- United States (20):
  - Arkansas Research Trials, LLC, North Little Rock, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Therapeutics Clinical Research, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Miami Dermatology and Laser Research, Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Medical Dermatology Specialists, Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Skin Sciences, Louisville, Kentucky
  - Derm Center, Troy, Michigan
  - ActivMed Practices and Research, Portsmouth, New Hampshire
  - Remington-Davis, Inc, Columbus, Ohio
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Paddington Testing Company Inc, Philadelphia, Pennsylvania
  - DermDox Centers for Dermatology, Sugarloaf, Pennsylvania
  - Studies in Dermatology, LLC, Cypress, Texas
  - Rodgers Dermatology, Frisco, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Complete Dermatology, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silverberg JI, Rosmarin D, Chovatiya R, Bieber T, Schleicher S, Beck L, Gooderham M, Chaudhry S, Fanton C, Yu D, Levy J, Liu Y, Miyazaki T, Tagliaferri M, Schmitz C, Nirula A, Kotzin B, Zalevsky J. The regulatory T cell-selective interleukin-2 receptor agonist rezpegaldesleukin in the treatment of inflammatory skin diseases: two randomized, double-blind, placebo-controlled phase 1b trials. Nat Commun. 2024 Oct 25;15(1):9230. doi: 10.1038/s41467-024-53384-1. PMID 39455575
- See also: A Study of LY3471851 in Participants With Eczema — https://trials.lillytrialguide.com/en-US/trial/3Ex7XDC7Soi22zSKKaGtrA